CLINICAL TRIAL: NCT03241550
Title: A Phase 1, Open-label, Multicenter, Non-comparative Pharmacokinetics and Safety Study of Intravenous and Oral Isavuconazonium Sulfate in Pediatric Patients
Brief Title: A Study of Intravenous and Oral Isavuconazonium Sulfate in Pediatric Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Collaborators: Basilea Pharmaceutica International Ltd (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9766-CL-0046
Record Dates: First submitted 2017-08-03; First posted 2017-08-07 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Hematological Malignancy
Keywords: invasive fungal disease; Cresemba®; Hematological malignancy; isavuconazonium sulfate; ASP9766; isavuconazole; pediatric population
MeSH Terms: conditions — Hematologic Neoplasms; Invasive Fungal Infections | interventions — isavuconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- isavuconazonium sulfate IV cohort 1: 1 to < 6 years of age (Experimental): Patients will receive an intravenous (IV) loading regimen of isavuconazonium sulfate, which consists of a dose every 8 hours (+/- 2 hours) on days 1 and 2, followed by once daily IV maintenance dosing for up to 26 additional days (for a maximum of 28 days of dosing).
  Interventions: Drug: isavuconazonium sulfate - intravenous
- isavuconazonium sulfate IV cohort 2: 6 to < 12 years of age (Experimental): Patients will receive an IV loading regimen of isavuconazonium sulfate, which consists of a dose every 8 hours (+/- 2 hours) on days 1 and 2, followed by once daily IV maintenance dosing for up to 26 additional days (for a maximum of 28 days of dosing).
  Interventions: Drug: isavuconazonium sulfate - intravenous
- isavuconazonium sulfate IV cohort 3: 12 to < 18 years of age (Experimental): Patients will receive an IV loading regimen of isavuconazonium sulfate, which consists of a dose every 8 hours (+/- 2 hours) on days 1 and 2, followed by once daily IV maintenance dosing for up to 26 additional days (for a maximum of 28 days of dosing).
  Interventions: Drug: isavuconazonium sulfate - intravenous
- isavuconazonium sulfate oral cohort 4: 6 to < 12 years of age (Experimental): Patients will receive a loading regimen of isavuconazonium sulfate by oral administration, comprising one dose every 8 hours (+/- 2 hours) on days 1 and 2 (a total of six doses), followed by once daily oral maintenance dosing for up to 26 additional days (for a maximum of 28 days of dosing).
  Interventions: Drug: isavuconazonium sulfate - oral
- isavuconazonium sulfate oral cohort 5: 12 to < 18 years of age (Experimental): Patients will receive a loading regimen of isavuconazonium sulfate by oral administration, comprising one dose every 8 hours (+/- 2 hours) on days 1 and 2 (a total of six doses), followed by once daily oral maintenance dosing for up to 26 additional days (for a maximum of 28 days of dosing).
  Interventions: Drug: isavuconazonium sulfate - oral

INTERVENTIONS:
Drug: isavuconazonium sulfate - intravenous — IV infusion
  Other Names: Cresemba®
  Arms: isavuconazonium sulfate IV cohort 1: 1 to < 6 years of age; isavuconazonium sulfate IV cohort 2: 6 to < 12 years of age; isavuconazonium sulfate IV cohort 3: 12 to < 18 years of age
Drug: isavuconazonium sulfate - oral — Oral
  Other Names: Cresemba®
  Arms: isavuconazonium sulfate oral cohort 4: 6 to < 12 years of age; isavuconazonium sulfate oral cohort 5: 12 to < 18 years of age

SUMMARY:
The purpose of the study is to evaluate the pharmacokinetics (PK), safety and tolerability of multiple doses of intravenous (IV) and oral isavuconazonium sulfate administered daily in pediatric patients. The PK data will be utilized to establish a pediatric population PK model of isavuconazole, the active moiety of isavuconazonium sulfate.

ELIGIBILITY:
Inclusion Criteria:

* Subject has sufficient venous access to permit administration of study drug (for the IV cohorts), collection of pharmacokinetic samples and monitoring of safety laboratories.
* Female subject must either:

  * Be of non-childbearing potential: Clearly premenarchal or documented surgically sterile
  * Or, if of childbearing potential: Agree not to try to become pregnant during the study and for 28 days after the final study drug administration; and have a negative urine or serum pregnancy test at screening; and, if heterosexually active, agree to consistently use 2 forms of highly effective birth control (at least one of which must be a barrier method) starting at screening and throughout the study and for 28 days after the final study drug administration.
* Female subject who is of childbearing potential must agree not to breastfeed starting at screening and throughout the study and for 28 days after the final study drug administration.
* Female subject who is of childbearing potential must not donate ova starting at screening and throughout the study and for 28 days after the final study drug administration.
* Male subject who is of childbearing potential and their female spouse/partner who is of childbearing potential must be using highly effective contraception consisting of 2 forms of birth control (at least one of which must be a barrier method) starting at screening and continue throughout the study, and for 90 days after the final study drug administration.
* Male subject who is of childbearing potential must not donate sperm starting at screening and throughout the study and, for 90 days after the final study drug administration.
* Subject and subject's parent(s) or legal guardian agree that the subject will not participate in another interventional study while on treatment.
* For oral cohorts: subject is able to swallow the oral capsule medication.

Exclusion Criteria:

* Subject has familial short QT syndrome, is receiving medications that are known to shorten the QT interval, or has a clinically significant abnormal electrocardiogram (ECG).
* Subject has evidence of hepatic dysfunction defined as:

  * Total bilirubin ≥ 3 times the upper limit of normal (ULN)
  * Alanine transaminase or aspartate transaminase ≥ 5 times the ULN
  * Known cirrhosis or chronic hepatic failure
* Subject has used strong cytochrome P450 (CYP) 3A4 inhibitors or inducers such as ketoconazole, rifampin/rifampicin, long acting barbiturates, carbamazepine and St. John's wort in the 5 days prior to the first administration of study drug.
* Subject has known history of allergy, hypersensitivity, or any serious reaction to any of the azole class antifungals.
* Subject has any condition which makes the subject unsuitable for study participation.
* Subject is unlikely to survive 30 days.
* Subject has received investigational therapy, with the exception of oncology drug trials, within 28 days or 5 half-lives, whichever is longer, prior to screening.
* For oral cohorts: The subject has gastrointestinal disease or has had a procedure that is expected to interfere with the oral absorption or tolerance of the study drug (e.g., functionally relevant gastrointestinal obstruction, mucositis/stomatitis, or frequent vomiting).
* Subject previously dosed with isavuconazonium sulfate.

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 49 (Actual)
Dates: Start 2017-10-02 (Actual); Primary Completion 2019-07-05 (Actual); Study Completion 2019-07-05 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK) of isavuconazole in plasma: Cmax at steady state | Up to 7 days
  Maximum concentration at steady state (Cmax) will be derived from the PK plasma samples collected.
PK of isavuconazole in plasma: AUCtau | Up to 7 days
  Area under the concentration time curve from the time of dosing to the start of next dosing interval at multiple dose conditions (AUCtau) will be derived from the PK plasma samples collected.
PK of isavuconazole in plasma: tmax | Up to 7 days
  Time of maximum concentration (tmax) will be derived from the PK plasma samples collected.
PK of isavuconazole in plasma: Ctrough | Up to 28 days
  Concentration - trough level (Ctrough) will be derived from the PK plasma samples collected.
PK of isavuconazole in plasma: CL | Up to 28 days
  Clearance (CL) will be model-derived.
PK of isavuconazole in plasma: Vss | Up to 28 days
  Volume of distribution at steady state (Vss) will be model-derived.
PK of isavuconazole in plasma: AUCss | Up to 28 days
  Area under the concentration-time curve at steady state (AUCss) will be model-derived.
PK of isavuconazole in plasma: t 1/2 | Up to 28 days
  Half-life (t1/2) will be model-derived.
Safety assessed by nature, frequency and severity of Treatment Emergent Adverse Events (TEAEs) | Up to 58 days
  A TEAE is defined as an Adverse Event (AE) observed after starting administration of the study drug through follow-up. AEs will be coded using the Medical Dictionary for Regulatory Activities (MedDRA). Number of patients with TEAE's will be summarized.
Number of patients with vital sign abnormalities and/or adverse events | Up to 28 days
  An abnormality identified during a medical test (e.g. vital signs) should be defined as an AE only if the abnormality meets 1 of the following criteria: induces clinical signs or symptoms; requires active intervention; requires interruption or discontinuation of study drug; or the abnormality or test value is clinically significant.
Number of patients with laboratory value abnormalities and/or adverse events | Up to 28 days
  An abnormality identified during a medical test (e.g. laboratory parameter) should be defined as an AE only if the abnormality meets 1 of the following criteria: induces clinical signs or symptoms; requires active intervention; requires interruption or discontinuation of study drug; or the abnormality or test value is clinically significant.
Safety assessed by routine 12- lead electrocardiogram (ECG) | Up to 28 days
  Standard 12-lead ECG recordings will be used for the purposes of safety assessment. A 12-lead, resting ECG is to be recorded. Patients should remain supine for at least 5 minutes prior to all ECGs being performed. The results (normal, abnormal not clinically significant, abnormal clinically significant) are to be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Senior Medical Director, Study Director — Astellas Pharma Global Development, Inc.
Locations (16):
- United States (16):
  - Miller Children's Hospital, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - CHOC Children's Hospital of Orange County, Orange, California
  - Nicklaus Children's Hospital, Miami, Florida
  - Emory University School of Medicine, Atlanta, Georgia
  - Ann & Robert H Lurie Children's Hospital of Chicago, Chicago, Illinois
  - University of Louisville, Louisville, Kentucky
  - Children's Hospitals and Clinics of Minnesota, Minneapolis, Minnesota
  - Children's Mercy Kansas City, Kansas City, Missouri
  - Duke University Medical Center, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - University Hospital of Cleveland, Cleveland, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - The Children's Hospital at TriStar Centennial Medical Center, Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Texas Children's Hospital, Houston, Texas

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- [Derived] Arrieta AC, Neely M, Day JC, Rheingold SR, Sue PK, Muller WJ, Danziger-Isakov LA, Chu J, Yildirim I, McComsey GA, Frangoul HA, Chen TK, Statler VA, Steinbach WJ, Yin DE, Hamed K, Jones ME, Lademacher C, Desai A, Micklus K, Phillips DL, Kovanda LL, Walsh TJ. Safety, Tolerability, and Population Pharmacokinetics of Intravenous and Oral Isavuconazonium Sulfate in Pediatric Patients. Antimicrob Agents Chemother. 2021 Jul 16;65(8):e0029021. doi: 10.1128/AAC.00290-21. Epub 2021 Jul 16. PMID 34031051
- See also: Link to results and other applicable study documents on the Astellas Clinical Trials website — https://www.clinicaltrials.astellas.com/study/9766-CL-0046/
- See also: Link to plain language summary of the study on the Trial Results Summaries website — https://www.trialsummaries.com/Study/StudyDetails?id=25654&tenant=MT_AST_9011